CLINICAL TRIAL: NCT04267991
Title: Corneal Densitometry Changes With Adenoviral Keratoconjunctivitis Sub Epithelial Infiltrates
Brief Title: Corneal Densitometry Changes With Adenoviral SEI
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Lecturer, Benha University
Other Study IDs: Hamaky5
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Corneal Disease
Keywords: adenoviral; infiltrates; PTK; tacrolimus
MeSH Terms: conditions — Corneal Diseases; Adenoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Tacrolimus: Patients were treated with 0.03 % tacrolimus ointment twice daily for 6 months.
  Interventions: Drug: Tacrolimus ointment
- Phototherapeutic Keratectomy: Patients underwent transepithelial PTK for subepithelial infiltrates.
  Interventions: Procedure: phototherapeutic keratectomy
- Control: patients received only artificial tears eyedrop

INTERVENTIONS:
Drug: Tacrolimus ointment — Patients were treated with 0.03 % tacrolimus ointment twice daily for 6 months.
  Other Names: Protopic ointment
  Groups: Tacrolimus
Procedure: phototherapeutic keratectomy — Patients underwent transepithelial PTK for subepithelial infiltrates.
  Groups: Phototherapeutic Keratectomy

SUMMARY:
Adenoviral Sub epithelial infiltrates (SEI) affect ocular function.They lead to reduced vision, photophobia, glare, halos, and foreign body sensation.

DETAILED DESCRIPTION:
first group of patients were treated with 0.03 % tacrolimus ointment twice daily for 6 months.S econd group underwent transepithelial PTK for subepithelial infiltrates. Baseline and post-treatment full ophthalmic examination was done.

ELIGIBILITY:
Inclusion Criteria:

* adenoviral SEI

Exclusion Criteria:

* Other corneal diseases

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 patients with adenoviral SEI
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
changes of corneal densitometry | 6 months
  Sub epithelial infiltrates was examined with the densitometry programme of the Pentacam (Fa. Oculus,Weimar, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: TAREK R ELHAMAKY, Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Elhamaky TR. Pentacam corneal densitometry-guided treatment of adenoviral corneal subepithelial infiltrates: a comparative study between transepithelial phototherapeutic keratectomy and topical tacrolimus. Int Ophthalmol. 2021 Jan;41(1):67-77. doi: 10.1007/s10792-020-01553-8. Epub 2020 Aug 27. PMID 32852646